CLINICAL TRIAL: NCT03961867
Title: S-1 Plus Docetaxel(DS) Versus S-1 Plus Oxaliplatin(SOX) as Postoperative Therapy for Stage II / III Gastric Cancer, a Randomized Controlled Trial
Brief Title: Docetaxel Versus Oxaliplatin as Addition to S-1 for Stage II / III Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Associate Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO203
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DS (Experimental): D2 resection -- S1 * 1 cycle + DS * 6 cycles + S1 * 9 cycles
  Interventions: Drug: Docetaxel
- SOX (Active Comparator): D2 resection -- SOX * 8 cycles + S1 * 8 cycles
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel — S-1 (BSA <1.25m2, 80 mg; 1.25 to 1.5m2, 100 mg; >1.5m2,120 mg) divided into two doses /day after breakfast and dinner, 14 days / 3 weeks, totally 16 cycles.
  Docetaxel 40mg/m2/3w from the second to the seventh cycles.
  Other Names: S-1
  Arms: DS
Drug: Oxaliplatin — S-1 (BSA <1.25m2, 80 mg; 1.25 to 1.5m2, 100 mg; >1.5m2,120 mg) divided into two doses /day after breakfast and dinner, 14 days / 3 weeks, totally 16 cycles.
  Oxaliplatin 130mg/m2/3w from the first to the eight cycles.
  Other Names: S-1
  Arms: SOX

SUMMARY:
S-1 plus oxaliplatin has been proved better than S-1 alone for stage II or III gastric cancer.

Docetaxel also showed excellent efficacy with S-1 in the postoperative setting for stage III gastric cancer.

This trial is designed to investigate the efficacy and safety of S-1 plus docetaxel versus S-1 plus oxalipltin as adjuvant chemotherapy after D2 resection in stage II / III gastric cancer.

DETAILED DESCRIPTION:
In this study, patients with gastric or EGJ adenocarcinoma who received D2 dissection and staged II or III, aged from 18 to 75 years and with ECOG PS ≤2 and adequate organ function, are stratified randomized according to pstage and location of primary lesion.

Group DS:

S-1 is orally administer by BSA (<1.25m2, 80 mg; 1.25 to 1.5m2, 100 mg; >1.5m2,120 mg) divided into two doses a day after breakfast and dinner for 14 days every three weeks to a total of 16 cycles postoperatively.

Docetaxel 40mg/m2/3w from the second to the seventh cycles.

Group SOX:

S-1 is orally administer by BSA (<1.25m2, 80 mg; 1.25 to 1.5m2, 100 mg; >1.5m2,120 mg) divided into two doses a day after breakfast and dinner for 14 days every three weeks to a total of 16 cycles postoperatively.

Oxaliplatin 130mg/m2/3w from the first to the eight cycles.

The primary end point is disease-free survival(DFS). The overall survival (OS), safty and quality of life are secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* informed consensus of patients
* be able to receive oral administration
* from 18 to 75 years old
* be proven to be primary adenocarcinoma of stomach and staged II or III by pathological evidences
* without other chemotherapy and/or radiation against to the disease
* normal function of other organs including heart,liver ,kidney and so on
* Eastern Cooperative Oncology Group performance status:0~2

Exclusion Criteria:

* history of other malignancy
* allergic reaction to S-1 or oxaliplatin of docetaxel
* be enrolling in other clinical trials
* abnormal GI tract function
* dysfunction of other organs
* female in pregnancy or lactation,or refuse to receive Contraception measures during chemotherapy
* other situation to be judged not adaptive to the study by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 year
  The interval from randomization to local recurrence, distant metastasis, death or the last follow-up

SECONDARY OUTCOMES:
overall survival | 5 year
  The interval from randomization to death or the last follow-up
Treatment related Adverse Events | 1 year
  According to CTC version 5

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No